CLINICAL TRIAL: NCT00681226
Title: ACE Inhibition; A Potential New Therapy for Peripheral Arterial Disease
Brief Title: Angiotensin Converting Enzyme (ACE) Inhibition and Peripheral Arterial Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayside Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 273/06
Record Dates: First submitted 2008-05-20; First posted 2008-05-21 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; angiotensin converting enzyme inhibitors; exercise
MeSH Terms: conditions — Peripheral Arterial Disease; Motor Activity | interventions — Ramipril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ramipril or matching placebo — 10 mg Ramipril or matching placebo once daily for 6 months
  Other Names: Ramace

SUMMARY:
Leg pain caused by peripheral arterial disease (PAD) can severely impede walking ability. Our preliminary findings indicate that the drug ramipril is much more effective in improving walking ability than current therapies. To be accepted as a new treatment for PAD these findings require validation in a much larger clinical trial.We propose to examine the effects of ramipril therapy for 6 months in a randomized, controlled trial of patients with PAD. If positive, this study will identify ramipril as a potential new therapy for PAD.

DETAILED DESCRIPTION:
This proposal extends our novel finding that the angiotensin-converting enzyme (ACE) inhibitor, ramipril markedly improves walking ability in patients with peripheral arterial disease (PAD), by conducting a larger clinical trial including a broader cross-section of PAD patients.

Hypothesis:

That ramipril therapy for 24 weeks will result in clinically significant increases in both pain-free and maximum walking time and improve quality of life in patients with PAD.

Background Synopsis:

Peripheral arterial disease is a common disorder, with 12% of adults over 50 having an ankle-brachial index (ABI) diagnostic of PAD (<0.9). Approximately one third of these patients experience intermittent claudication during walking, limiting the ability of these older individuals to participate in normal activities. The aim of PAD treatment is to improve walking distance and quality of life in those with intermittent claudication, and to decrease long term cardiovascular morbidity and mortality. However, the range of medical treatments to improve walking distance in these patients is limited. Our pilot study demonstrates that treatment of PAD patients, with infra-inguinal disease and without diabetes with ramipril for 24 weeks, markedly improves waking ability. Relative to placebo, ramipril increased mean treadmill-assessed pain-free waking time by 227s (160%, p<0.001) and mean maximum walking time by 451s (240%, p<0.001). Assuming a constant speed of 0.89 m/s (3.2 km/hr), this corresponds to a clinically significant increase in walking distance of 401m (95% CI 330m to 480m) which would impact appreciably on daily functional capacity. The magnitude of this effect is significantly greater than that reported for conventional medical therapies and provides worthwhile clinical benefit.

Research Plan Synopsis:

The dramatic findings of our pilot study clearly warrant verification in a larger clinical trial including diabetic patients and those with aorto-iliac disease as well as infra-inguinal disease. The current proposal is to expand our pilot study into a large trial with broad inclusion criteria. We propose to include patients with diabetes mellitus not currently medicated with ACE inhibitors. 264 PAD patients will be randomised to either ramipril (10mg once daily) or matching placebo for 24 weeks in a randomised, double-blind placebo controlled trial. All patients will undergo a treadmill exercise test to determine pain free and maximum walking times, ABI measurements and Duplex scanning to determine stenosis severity, both at baseline and following 6 months of ramipril therapy. Functional capacity in a daily life setting, will be assessed using standardised questionnaires (Walking Impairment Questionnaire and Quality of Life Questionnaire).

Outcomes and Significance:

If positive this trial will validate our pilot findings that the ACE inhibitor ramipril is an efficacious new therapy for the treatment of patients with claudication resulting from PAD. Given the escalating prevalence of PAD, this work has the potential for widespread impact.

ELIGIBILITY:
Inclusion Criteria:

* Ankle brachial index of <0.9 in at least one leg
* History of intermittent claudication (unilateral or bilateral)
* A stable medication regimen for at least 6 months

Exclusion Criteria:

* Limiting coronary artery disease
* Renal failure (serum creatinine > 0.20 mmol/L)
* Current treatment or treatment within the previous 6 months with ACE inhibitors or angiotensin II receptor antagonists

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-01; Primary Completion 2011-08 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
walking time | baseline and 6 months

SECONDARY OUTCOMES:
walking impairment questionnaire | baseline and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn A Kingwell, PhD, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Baker Heart Research Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Background] Ahimastos AA, Lawler A, Reid CM, Blombery PA, Kingwell BA. Brief communication: ramipril markedly improves walking ability in patients with peripheral arterial disease: a randomized trial. Ann Intern Med. 2006 May 2;144(9):660-4. doi: 10.7326/0003-4819-144-9-200605020-00009. PMID 16670135 (Retraction: PMID 26544086 Ann Intern Med. 2015 Dec 1;163(11):884)
- [Derived] Ahimastos AA, Latouche C, Natoli AK, Reddy-luthmoodoo M, Golledge J, Kingwell BA. Potential vascular mechanisms of ramipril induced increases in walking ability in patients with intermittent claudication. Circ Res. 2014 Mar 28;114(7):1144-55. doi: 10.1161/CIRCRESAHA.114.302420. Epub 2014 Jan 7. PMID 24397981 (Retraction: PMID 26358112 Circ Res. 2015 Sep 11;117(7):e64)
- [Derived] Ahimastos AA, Walker PJ, Askew C, Leicht A, Pappas E, Blombery P, Reid CM, Golledge J, Kingwell BA. Effect of ramipril on walking times and quality of life among patients with peripheral artery disease and intermittent claudication: a randomized controlled trial. JAMA. 2013 Feb 6;309(5):453-60. doi: 10.1001/jama.2012.216237. PMID 23385271 (Retraction: PMID 26367349 JAMA. 2015 Oct 13;314(14):1520-1)